CLINICAL TRIAL: NCT00056381
Title: Phase I/II Study of the Safety, Tolerance and Pharmacokinetics of Anidulafungin in Immunocompromised Children With Fever and Neutropenia
Brief Title: Safety, Tolerance and Pharmacokinetics of Anidulafungin in Immunocompromised Children Ages 2-17
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Vicuron Pharmaceuticals (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VER002-12; A8851005
Record Dates: First submitted 2003-03-11; First posted 2003-03-12 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Neutropenia
Keywords: neutropenia; fever; febrile neutropenia
MeSH Terms: conditions — Neutropenia; Fever; Febrile Neutropenia | interventions — Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin

SUMMARY:
Anidulafungin is a medicine being developed for treatment of adults with certain kinds of fungal infections. This study is evaluating anidulafungin in children and adolescents who have fever and a low white blood cell count (neutropenia).

DETAILED DESCRIPTION:
Anidulafungin is an investigational drug being developed as an intravenous treatment for esophageal candidiasis, candidemia and other invasive fungal infections. Anidulafungin is an antifungal agent of the echinocandin class, which targets the fungal cell wall of yeast and other filamentous fungi.

ELIGIBILITY:
* Children ages 2-17 years with fever and neutropenia.
* The expected duration of neutropenia should be 10 days and due to cytotoxic chemotherapy or aplastic anemia.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2003-07; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Versicor, King of Prussia, Pennsylvania, United States